CLINICAL TRIAL: NCT03434184
Title: Observational Prospective Comparative Study Before and After Spinal Surgery for Scoliosis With Pelvic Fixation in Patients
Brief Title: Study of Walk in Patients With Pelvic Fixation
Acronym: FBPM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI17021J; 2017-A02486-47 (Other: ID-RCB)
Record Dates: First submitted 2018-01-24; First posted 2018-02-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis
Keywords: Walking analysis; spinal surgery; scoliosis; pelvic fixation
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to determine the effect of double end spinal instrumentation from the upper thoracic to the pelvis with sacro-iliac ﬁxation on the gait of ambulating patients with pelvic obliquity 6 month after surgery.

DETAILED DESCRIPTION:
The pelvic fixations were used since many years for these patients. However there are no prospective study investigating the gait evolution before and after a surgical treatment by long spinal instrumentation with pelvic fixation.

Investigators are planning to analyze the gait, before and 6 months after surgery. Investigators will use 2 qualitative criterions with a gait analysis and a walking test, and 1 quantitative criterion with a questionnaire assessing the patient's functional change. Investigators will use as surgical treatment a long double end spinal fixation without fusion, investigators use an ilio sacral screw as pelvic anchor on each side.

Evaluation of changes in gait after pelvic fixation of a long spinal instrumentation will make it possible to extend or, on the contrary, restrict the indications for pelvic fixation surgery in walking patients, who are candidates for pelvic fixation.

ELIGIBILITY:
Inclusion Criteria:

* Patient under 18 walking or strolling
* Patient with scoliosis requiring long instrumentation taking pelvis with iliosacral screws

Exclusion Criteria:

* Patient presenting a predictable pejorative evolution of the walk due to the pathology of the patient within 2 years
* Patient or parent who has notified their refusal to participate

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under 18 years of age who are walking requiring spinal instrumentation taking the pelvis taken care of in the orthopedic department of NECKER.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Change in the score of CPCHILD (section 2) questionnaire from 6 months before spinal surgery at 6 month after spinal surgery | 6 months before and 6 months after spinal surgery
  to assess the quality criteria of walk
Change in Clinical Gait Analysis from 6 months before spinal surgery at 6 month after spinal surgery | 6 months before and 6 months after spinal surgery
  to assess the quantitative criteria of walk
Change in 6-minute walking test from 6 months before spinal surgery at 6 month after spinal surgery | 6 months before and 6 months after spinal surgery
  to assess the quantitative criteria of walk

SECONDARY OUTCOMES:
presence / absence of cardiac impairment | 6 months before spinal surgery
  cardiac evaluation to evaluate assess if cardiac impairment before spinal surgery is a the good or bad prognosis for walking
presence / absence of respiratory impairment | 6 months before spinal surgery
  pulmonary evaluation to assess if respiratory impairment before spinal surgery is a good or bad prognosis for walking
presence / absence of neurological impairment | 6 months before spinal surgery
  neurological evaluation to assess if neurology impairment before spinal surgery is a good or bad prognosis for walking
Change in reducibility of scoliosis from 6 months before spinal surgery at 6 month after spinal surgery | 6 months before and 6 months after spinal surgery
  to evaluate the good or bad prognosis for walking
Change in "holding of the head " of scoliosis : from 6 months before spinal surgery at 6 month after spinal surgery | 6 months before and 6 months after spinal surgery
  to evaluate the good or bad prognosis for walking
Change in curvature of scoliosis from 6 months before spinal surgery at 6 month after spinal surgery | 6 months before and 6 months after spinal surgery
  to evaluate the good or bad prognosis for walking
Change in imbalance of scoliosis from 6 months before spinal surgery at 6 month after spinal surgery | 6 months before and 6 months after spinal surgery
  to evaluate the good or bad prognosis for walking

CONTACTS AND LOCATIONS:
Overall Officials: Lotfi MILADI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No